CLINICAL TRIAL: NCT02983383
Title: Effect of TAP Block for Postoperative Pain Control After Varicocele Operations on Analgesia Quality and Postoperative Analgesic Consumption
Brief Title: Effect of TAP Block for Postoperative Pain Control After Varicocele Operations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Boran, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 53
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Varicocele
Keywords: Varicocele; TAP block; spinal anesthesia
MeSH Terms: conditions — Varicocele | interventions — Sensitivity Training Groups; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP block group (Group T) (Active Comparator): At the end of the operation, patients in Group T in the supine position will have a USI probe placed at the middle point between the costal edge and iliac crest (within the Petit triangle) after necessary antiseptic conditions are ensured. Then after the abdominal muscle layers are observed, the needle tip will be advanced through the muscle layers and pass the fascia, feeling the fascial click, monitored by USI in controlled fashion. After feeling the second click (passing the internal oblique muscle fascia), a test dose of 0.5-1 ml saline will be administered to determine the localization of the needle tip. Then noting the location, with frequent aspiration local anesthetic agent will be administered to the neurofascial plane for TAP block.
  Interventions: Procedure: TAP block group (Group T)
- Group without TAP (Group P) (Active Comparator): Patients in Group P will have adjuvant added to spinal anesthesia.
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: TAP block group (Group T) — At the end of the operation, patients in Group T in the supine position will have a USI probe placed at the middle point between the costal edge and iliac crest (within the Petit triangle) after necessary antiseptic conditions are ensured. Then after the abdominal muscle layers are observed, the needle (Stimuplex Ultra 22G, 100mm, B.Braun, Germany) tip will be advanced through the muscle layers and pass the fascia, feeling the fascial click, monitored by USI in controlled fashion. After feeling the second click (passing the internal oblique muscle fascia), a test dose of 0.5-1 ml saline will be administered to determine the localization of the needle tip. Then noting the location, with frequent aspiration local anesthetic agent will be administered to the neurofascial plane for TAP block.
  Arms: TAP block group (Group T)
Procedure: spinal anesthesia — Patients in Group P will have adjuvant added to spinal anesthesia (25 G, Quincke spinal anesthesia needle, Egemen,Turkey).
  Arms: Group without TAP (Group P)

SUMMARY:
TAP block is the administration of local anesthetic agents into the anatomic neurofascial cavity between the internal oblique and transversus abdominis muscle in the antero-lateral region of the abdomen to block the anterior branches of the thoracic intercostal (T7-T12) and first lumbar (L1) nerves. TAP block may be a good method for postoperative pain control. We aim to show the effect of TAP block administration on analgesic consumption after varicocelectomy operations, side effects linked to analgesic use and analgesic quality.

DETAILED DESCRIPTION:
The study will include 50 patients aged from 18-45 years in ASA I-II risk group undergoing varicocelectomy operations under elective conditions, randomized with a lottery method. Patients will be informed of the study and included in the study after giving permission with a patient consent form. Patients will be divided into two groups; TAP group (Group T, n=25) and P (Group P, n=25). Both groups will be taken for operation under spinal anesthesia. Those with contraindications for spinal anesthesia, with coagulopathy, with known allergy to the medications used, with infection in the operated area, and those who do not volunteer will be excluded from the study. At the end of the operation, patients in Group T in the supine position will have a USI probe placed at the middle point between the costal edge and iliac crest (within the Petit triangle) after necessary antiseptic conditions are ensured. Then after the abdominal muscle layers are observed, the needle tip will be advanced through the muscle layers and pass the fascia, feeling the fascial click, monitored by USI in controlled fashion. After feeling the second click (passing the internal oblique muscle fascia), a test dose of 0.5-1 ml saline will be administered to determine the localization of the needle tip. Then noting the location, with frequent aspiration local anesthetic agent will be administered to the neurofascial plane for TAP block. Patients in Group P will have adjuvant added to spinal anesthesia. Patients in both groups will have pain scores assessed at 2, 4, 6, 12 and 24 hours postoperative at rest and coughing with VAS (visual analog scale) (pain severity: 0 no pain to 10 most severe pain experienced to date) and values will be recorded. When patients are in pain, analgesic agent will be administered according to patient controlled analgesia protocol. The time of first requirement for analgesic agent and the amount of analgesic agent used in 24 hours will be recorded for patients. Side effects like postoperative nausea, vomiting, or itching will be noted. Additionally, patient satisfaction will be assessed by asking if the surgical method they experienced was bad, moderate, good or very good and recorded.

ELIGIBILITY:
Inclusion Criteria:

18-45 year old ASA I-II patient group

Exclusion Criteria:

1. Contraindications for spinal anesthesia
2. Coagulopathy
3. Known allergy to medications used
4. Infection in the operated area
5. Non-volunteer patient

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
VAS (visual analog scale) | 24 Hours
  VAS (visual analog scale) (pain severity: 0 no pain to 10 most severe pain experienced to date) score changes in the postoperative period at rest and coughing
Postoperative side effects | 24 Hours
  questionnaire for postoperative nausea, vomiting, numbness and itching
Patient satisfaction | 24 Hours
  questionnaire for patient satisfaction
time to first analgesic | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Faruk Boran, Study Chair — Kahramanmaraş Üniversitesi
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No